CLINICAL TRIAL: NCT01225627
Title: Effects of Discharge Coordinator Intervention on Hospitalizations and Quality of Life in Patients With Chronic Obstructive Pulmonary Disease: a Randomized Controlled Clinical Trial
Brief Title: Discharge Coordinator Intervention in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University Clinic of Pulmonary and Allergic Diseases Golnik (Other)
Responsible Party: Principal Investigator, Mitja Lainščak, Professor, The University Clinic of Pulmonary and Allergic Diseases Golnik
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Golnik-COPD-DC-1
Record Dates: First submitted 2010-10-18; First posted 2010-10-21 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic disease management; Chronic obstructive pulmonary disease; Discharge planning; Discharge coordinator
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coordinated discharge (Experimental): Patients will receive support by discharge coordinator for activities associated with discharge and immediate post-discharge care.
  Interventions: Other: Coordinated discharge
- Control (Placebo Comparator): Patients in control group will be managed by attending physician, primary care physician, and/or pneumologist in accordance with established clinical practice.
  Interventions: Other: Control

INTERVENTIONS:
Other: Coordinated discharge — In intervention group, a discharge coordinator contacts hospitalized patients the day after randomization. During hospitalization, discharge coordinator visits are scheduled according to patients' problems and home-care needs. At 48 hours after hospital discharge, a discharge coordinator calls patients by phone to check the process of adjustment to home environment and to inquire about additional needs patients might have. Thereafter, phone contacts are scheduled according to the patients' needs and 7-10 days after the hospital discharge a home visit is performed by discharge coordinator, respectively.
  Arms: Coordinated discharge
Other: Control — Patients in control group will be managed by attending physician, primary care physician, and/or pneumologist in accordance with established clinical practice.
  Arms: Control

SUMMARY:
This is a single-centre randomized controlled clinical trial which will enroll COPD patients in Global Initiative for Chronic Obstructive Lung Disease (GOLD) stage II-IV, hospitalized due to acute exacerbation. Patients will be randomised in a 1:1 fashion to intervention group, which will have care organized by discharge coordinator, and control group which will receive care as usual. The primary endpoint of this study is time to hospitalization due to COPD worsening. Data will be collected at baseline, at the time of hospital discharge, and at following time-points after the hospital discharge: 48 hours, 7-10 days, 30 days, 90 days, and 180 days.

DETAILED DESCRIPTION:
This is a single-centre randomized controlled clinical trial to assess the effectiveness of discharge coordinator intervention compared to care as usual in patients with COPD.

The study is being conducted at University Clinic of Pulmonary and Allergic Diseases Golnik, Slovenia. Patients with suspicion of acute exacerbation of COPD will be screened at admission when they will be informed about study details. After explanations of concerns and questions that they might have, a signed informed consent will be collected. During 48 hours, patients will be included according to their eligibility. Main inclusion criteria are COPD stage II-IV according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines, ability to perform phone contacts and availability for home visits. Patients will be excluded if in unstable or terminal stage of disease other than COPD, if they will die during hospitalization, or if unable to follow the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* age >35 years
* acute exacerbation of COPD stage II-IV
* residence in the geographical area linked to the study hospital
* ability to communicate
* give written informed consent

Exclusion Criteria:

* diagnosis of cognitive impairment
* unstable or terminal disease other than COPD
* withdrawal of written informed consent before discharge
* inability of phone contact
* death during hospitalisation

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2009-11; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Number of patients hospitalized due to COPD worsening | 180 days
  A hospitalization is defined as an unplanned overnight stay in hospital (different date for admission and discharge) due to acute worsening of COPD. Endpoint will be adjudicated by Endpoint committee.

SECONDARY OUTCOMES:
All-cause mortality | 180 days
  Mortality will be ascertained at the Central Population Registry.
Acute exacerbations of COPD | 180 days
  Endpoint will be adjudicated by Endpoint committee.
Time to hospitalization due to COPD worsening | 180 days
  A hospitalization is defined as an unplanned overnight stay in hospital (different date for admission and discharge) due to acute worsening of COPD. Endpoint will be adjudicated by Endpoint committee.
Days alive and out of hospital | 180 days
  Endpoint will be adjudicated by Endpoint committee.
Health-related quality of life | 180 days
  Endpoint will be adjudicated by Endpoint committee.
Health care costs | 180 days
  Endpoint will be adjudicated by Endpoint committee.

CONTACTS AND LOCATIONS:
Overall Officials: Mitja Lainscak, MD, PhD, Study Chair — University Clinic Golnik; Jerneja Farkas, MD, PhD, Principal Investigator — University of Ljubljana
Locations (1):
- University Clinic Golnik, Golnik, Slovenia

REFERENCES:
- [Background] Farkas J, Kadivec S, Kosnik M, Lainscak M. Effectiveness of discharge-coordinator intervention in patients with chronic obstructive pulmonary disease: study protocol of a randomized controlled clinical trial. Respir Med. 2011 Oct;105 Suppl 1:S26-30. doi: 10.1016/S0954-6111(11)70007-5. PMID 22015082